CLINICAL TRIAL: NCT03403712
Title: A Multicenter, Randomized, Double-blind, Double-dummy, Active-controlled, Parallel Group Phase 3b Study to Assess the Safety and to Describe the Efficacy of IV Fosnetupitant/Palonosetron (260 mg/0.25 mg) Combination (IV NEPA FDC) Compared to Oral Netupitant/Palonosetron (300 mg/0.5 mg) Combination (Akynzeo®) for the Prevention of Chemotherapy-induced Nausea and Vomiting in Initial and Repeated Cycles of Anthracycline-cyclophosphamide (AC) Chemotherapy in Women With Breast Cancer
Brief Title: A Study to Assess the Safety and the Efficacy of IV Fosnetupitant/Palonosetron (260 mg/0.25 mg) Combination Compared to Oral Netupitant/Palonosetron (300 mg/0.5 mg) Combination for the Prevention of CINV in AC Chemotherapy in Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Emerald Clinical Inc. (Industry); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NEPA-17-05
Record Dates: First submitted 2018-01-04; First posted 2018-01-19 (Actual); Results first posted 2020-04-15 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — netupitant, palosentron drug combination; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): intravenous fosnetupitant/ palonosetron (260 mg/0.25 mg) fixed-dose combination, administered as a 30-minute infusion of a 50 mL solution, on Day 1 of each cycle.
  Oral dexamethasone will be administered on Day 1 of each cycle (12 mg)
  Interventions: Drug: fosnetupitant/ palonosetron; Drug: dexamethasone
- Control group (Active Comparator): oral netupitant/palonosetron (300 mg/0.50 mg) fixed-dose combination on Day 1 of each cycle.
  Oral dexamethasone will be administered on Day 1 of each cycle (12 mg)
  Interventions: Drug: netupitant/palonosetron; Drug: dexamethasone

INTERVENTIONS:
Drug: fosnetupitant/ palonosetron — intravenous fosnetupitant/ palonosetron (260 mg/0.25 mg) fixed-dose combination
  Other Names: IV NEPA FDC
  Arms: Test group
Drug: netupitant/palonosetron — oral netupitant/palonosetron (300 mg/0.50 mg) fixed-dose combination
  Other Names: Akynzeo capsules
  Arms: Control group
Drug: dexamethasone — Oral dexamethasone (12 mg)

SUMMARY:
Multicenter, randomized, double-blind, double-dummy, parallel group, stratified study assessing the safety and describing the efficacy of a single dose of intravenous (IV) fosnetupitant/palonosetron (260 mg/0.25 mg) infusion [test] versus oral netupitant/palonosetron (300 mg/0.5 mg) combination [control]; each administered with oral dexamethasone prior to initial and repeated cycles of AC chemotherapy in female breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Cycle 1:

The following inclusion criteria must be checked prior to inclusion at Cycle 1:

1. Patient read, understood and signed the written informed consent before any study related activity, agreeing to participate in the study and to comply with study requirements.
2. Female patient of at least 8 years of age.
3. Histologically or cytologically confirmed breast cancer, including recurrent or metastatic.
4. Naïve to moderately or highly emetogenic antineoplastic agents.
5. Scheduled to receive at least 4 consecutive cycles of an AC combination regimen.

   Notes:
   1. additional not emetogenic, minimally or low emetogenic antineoplastic agents are permitted at any time after start of AC combination on Day 1.
   2. additional highly or moderately emetogenic antineoplastic agents are only allowed on Day 1 after the start of AC combination, provided their administration is completed within 6 hours from the start of the AC combination administration.
6. ECOG Performance Status of 0 or 1.
7. Patient shall be: a) of non-childbearing potential or b) of childbearing potential using reliable contraceptive measures and having a negative urine pregnancy test within 24 hours prior to dose of investigational product.

   Notes:
   1. Female patients of non-childberaring potential are defined as being in post-menopausal state since at least 1 year; or having documented surgical sterilization or hysterectomy at least 3 months before study participation.
   2. Reliable contraceptive measures include implants, injectables, combined oral contraceptives, intrauterine devices, vasectomized partner or complete (long term) sexual abstinence;
8. Hematologic and metabolic status adequate for receiving a cycle of AC chemotherapy based on investigator's assessment.
9. If the patient has a known hepatic or renal impairment, she may be enrolled in the study at the discretion of the Investigator.
10. Able to read, understand, follow the study procedure and complete the patient diary.

All inclusion criteria will be checked at screening visit (Visit 1 of Cycle 1); inclusion criteria 7 will be re-checked at Day 1 (Visit 2).

Cycles 2 to 4:

The following inclusion criteria must be checked prior to inclusion at each repeated cycle:

1. Participation in the study during the next cycle of chemotherapy is considered appropriate by the Investigator and does not pose unwarranted risk to the patient.
2. Scheduled to receive an AC chemotherapy regimen or AC chemotherapy together with other chemotherapies as defined in Inclusion criterion #5 for Cycle 1.
3. Patient shall be: a) of non-childbearing potential or b) of childbearing potential using reliable contraceptive measures and having a negative urine pregnancy test within 24 hours prior to dosing of investigational product.
4. Adequate hematologic and metabolic status for receiving a cycle of AC chemotherapy according to the Investigator's opinion.

All inclusion criteria will be checked at screening visit (Visit 1); inclusion criterion #3 will be re-checked at Day 1 (Visit 2).

Exclusion Criteria:

Cycle 1:

The following exclusion criteria must be checked prior to inclusion at Cycle 1:

1. Lactating patient.
2. Current use of illicit drugs or current evidence of alcohol abuse.
3. Scheduled to receive moderately or highly emetogenic antineoplastic agent in addition to the AC regimen, from 6 hours after the start of the AC chemotherapy on Day 1 and up to Day 1 of Cycle 2.
4. Received or is scheduled to receive radiation therapy to the abdomen or the pelvis within 1 week prior to the start of AC chemotherapy administration on Day 1 or between Days 1 to 5, inclusive.
5. Any vomiting, retching, or nausea (grade 1 as defined by National Cancer Institute) within 24 hours prior to the start of AC chemotherapy administration on Day 1.
6. Symptomatic primary or metastatic central nervous system (CNS) malignancy.
7. Active peptic ulcer disease, gastrointestinal obstruction, increased intracranial pressure, hypercalcemia, an active infection or any illness or medical conditions (other than malignancy) that, in the opinion of the Investigator, may confound the results of the study, represent another potential etiology for emesis and nausea (other than chemotherapy-induced nausea and vomiting [CINV]) or pose unwarranted risks in administering the study drugs to the patient.
8. Known hypersensitivity or contraindication to 5 hydroxytryptamine type 3 (5-HT3) receptor antagonists (e.g., palonosetron, ondansetron, granisetron, dolasetron, tropisetron, ramosetron), to dexamethasone, or to neurokinin-1 (NK1) receptor antagonists (e.g., aprepitant, rolapitant).
9. Known contraindication to the IV administration of 50 mL 5% glucose solution.
10. Participation in a previous clinical trial involving IV fosnetupitant or oral netupitant administered alone or in combination with palonosetron.
11. Any investigational drugs taken within 4 weeks prior to Day 1, and/or is scheduled to receive any investigational drug (other than those planned by the study protocol) during the present study.
12. Systemic corticosteroid therapy within 72 hours prior to the start of AC chemotherapy administration on Day 1, except the dexamethasone provided as additional study drug. However, topical and inhaled corticosteroids are permitted.
13. Scheduled to receive bone marrow transplantation and/or stem cell rescue therapy during the study participation.
14. Other than as administered as part of the study protocol, any medication with known or potential antiemetic activity within 24 hours prior to the start of AC chemotherapy administration on Day 1, including:

    * 5-HT3 receptor antagonists (e.g., ondansetron, granisetron, dolasetron, tropisetron, ramosetron, palonosetron)
    * NK1 receptor antagonists (e.g., aprepitant, fosaprepitant, rolapitant or any other new drug of this class)
    * benzamides (e.g., metoclopramide, alizapride)
    * phenothiazines (e.g., prochlorperazine, promethazine, fluphenazine, perphenazine, thiethylperazine, chlorpromazine)
    * benzodiazepines (except if the subject is receiving such medication for sleep or anxiety and has been on a stable dose for at least seven days prior to Day 1).
    * butyrophenones (e.g., haloperidol, droperidol)
    * anticholinergics (e.g., scopolamine, with the exception of inhaled anticholinergics for respiratory disorders, e.g., ipratropium bromide)
    * antihistamines (e.g., cyclizine, hydroxyzine, diphenhydramine, chlorpheniramine)
    * domperidone
    * mirtazapine
    * olanzapine
    * prescribed cannabinoids (e.g., tetrahydrocannabinol or nabilone)
    * Over The Counter (OTC) antiemetics, OTC cold or OTC allergy medications.
15. Scheduled to receive any strong or moderate inhibitor of CYP3A4 during the efficacy assessment period (Day 1 to Day 5, inclusive) or its intake within 1 week prior to Day 1.
16. Scheduled to receive any CYP3A4 inducer during the efficacy assessment period (Day 1 to Day 5, inclusive) or its intake within 4 weeks prior to Day 1, with the exception of corticosteroids (for which exclusion criterion #12 applies).
17. History or predisposition to cardiac conduction abnormalities, except for incomplete right bundle branch block.
18. History of risk factors for Torsades de Pointes (heart failure, hypokalemia, family history of Long QT Syndrome).
19. Severe or uncontrolled cardiovascular diseases, including myocardial infarction within 3 months prior to Day 1, unstable angina pectoris, significant valvular or pericardial disease, history of ventricular tachycardia, symptomatic Congestive Heart Failure (CHF) New York Heart Association (NYHA) class III-IV, and severe uncontrolled arterial hypertension.

All exclusion criteria with the exception of criteria #5, #12, and #14 will be checked at screening visit (Visit 1). Exclusion criteria #5, #12, and #14 will be checked at Day 1 (Visit 2) only.

Exclusion criteria #3, #4, #7, #11, #13, #15, and #16 need to be re-checked at Day 1 (Visit 2).

Cycles 2 to 4:

The following exclusion criteria must be checked prior to inclusion at each repeated cycle:

1. Scheduled to receive moderately or highly emetogenic antineoplastic agent in addition to the AC regimen, from 6 hours after the start of the AC chemotherapy on Day 1 of current cycle and up to Day 1 of the next cycle.
2. Active infection or uncontrolled disease that may pose unwarranted risks in administering the study drugs to the patient.
3. Started any of the prohibited medications.
4. Any vomiting, retching, or nausea (grade ≥ 1 as defined by National Cancer Institute) within 24 hours prior to the start of AC chemotherapy administration on Day 1.
5. Received or is scheduled to receive radiation therapy to the abdomen or the pelvis within 1 week prior to the start of AC chemotherapy administration on Day 1 or between Days 1 to 5.
6. Symptomatic primary or metastatic CNS malignancy.
7. Any illness or medical condition that, in the opinion of the investigator, may confound the results of the study or pose unwarranted risks in administering the investigational product or dexamethasone to the patient.

All exclusion criteria, with exception of criterion #4, will be checked at screening visit (Visit 1). Exclusion criterion #4 will be checked at Day 1 (Visit 2) only. Exclusion criteria #2, #3 and #5 need to be re-checked at Day 1 (Visit 2).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (36):
  - The Oncology Inst. Of Hope and Innovation, Tucson, Arizona
  - Carti Cancer Center, Little Rock, Arkansas
  - Pacific Cancer Medical Center, Inc., Anaheim, California
  - CBCC Global Research, INC at Comprehensive Blood and Cancer Center, Bakersfield, California
  - The Oncology Tnstitute of Hope and Innovation, Corona, California
  - Uptimum Medical Group Inc., Inglewood, California
  - The Oncology Institute of Hope and Innnovation, Long Beach, California
  - Hao Wei Zhang M.D., Los Angeles, California
  - Emad Ibrahim, MD, INC., Redlands, California
  - Watson Clinic LLP, Lakeland, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Cancer Center of !!Iiddle Georgia, Dublin, Georgia
  - Harbin Clinic, Rome, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - Edward H. Kaplan MD & Associates, Skokie, Illinois
  - Presence Infusion Care - Skokie, Skokie, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - TU Health Arnett Cancer Center, Lafayette, Indiana
  - Baptist Health Cancer Center, New Albany, Indiana
  - Cotton O'Neil Clinical Res. Ctr., Hematology & Oncology, Topeka, Kansas
  - Cancer Center of Kansas, Wichita, Kansas
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - CHRISTUS Cancer Treatment Center, Shreveport, Louisiana
  - Mercy Medical Center, Medical Oncology and Hematology, Baltimore, Maryland
  - Hattiesburg Clinic Hematology Oncology, Hattiesburg, Mississippi
  - Cornell-Beshore Cancer Institute, Joplin, Missouri
  - Cox Mcdical ·Centers, Springfield, Missouri
  - Trinitas Cancer Center, Elizabeth, New Jersey
  - San Juan Oncology Associates, Farmington, New Mexico
  - Mid Ohio Oncology/Hematology Inc. DBA The Mark H. Zangmeister Center, Columbus, Ohio
  - Toledo Clinic Cancer Center - Toledo, Toledo, Ohio
  - Monongahela Valley Hospital, Monongahela, Pennsylvania
  - Carolina Blood and Cancer Care Associates, P.A., Rock Hill, South Carolina
  - The West Clinic, PC dba West Cancer Center, Germantown, Tennessee
  - Cheyenne Regional Medical Center, Cheyenne, Wyoming
- Georgia (4):
  - JSC Saint Nikolozi Surgery and Oncological Centre, Kutaisi
  - LTD Institute of Clinical Oncology, Tbilisi
  - LTD Tbilisi Oncology Dispensary, Tbilisi
  - LTD S.Khechinashvili University Hospital, Tbilisi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Navari R, Binder G, Molasiotis A, Herrstedt J, Roeland EJ, Ruddy KJ, LeBlanc TW, Kloth DD, Klute KA, Papademetriou E, Schmerold L, Schwartzberg L. Duration of Chemotherapy-Induced Nausea and Vomiting (CINV) as a Predictor of Recurrent CINV in Later Cycles. Oncologist. 2023 Mar 17;28(3):208-213. doi: 10.1093/oncolo/oyac240. PMID 36527702

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 202 patients were randomized to IV NEPA and 202 patients were randomized to Oral NEPA. Two randomized patients (Patient IDs 211003 and 213001) in the IV NEPA group did not receive any active study drug or AC chemotherapy.
Groups:
- Test Group: intravenous fosnetupitant/ palonosetron (260 mg/0.25 mg) fixed-dose combination, administered as a 30-minute infusion of a 50 mL solution, on Day 1 of each cycle.
  Oral dexamethasone will be administered on Day 1 of each cycle (12 mg)
  fosnetupitant/ palonosetron: intravenous fosnetupitant/ palonosetron (260 mg/0.25 mg) fixed-dose combination
  dexamethasone: Oral dexamethasone (12 mg)
- Control Group: oral netupitant/palonosetron (300 mg/0.50 mg) fixed-dose combination on Day 1 of each cycle.
  Oral dexamethasone will be administered on Day 1 of each cycle (12 mg)
  netupitant/palonosetron: oral netupitant/palonosetron (300 mg/0.50 mg) fixed-dose combination
  dexamethasone: Oral dexamethasone (12 mg)
Period: Overall Study
Arm/Group | Test Group | Control Group
Started | 200 | 202
Completed | 95 | 102
Not Completed | 105 | 100

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test Group | Control Group | Total
Number analyzed (Participants) | 200 | 202 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.94) | 55.2 (9.73) | 55.4 (9.82)
Age, Customized [Count of Participants; unit: Participants]
  <55 years | 89 | 91 | 180
  >55 years | 111 | 111 | 222
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 202 | 402
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 192 | 189 | 381
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 9 | 13
  White | 189 | 186 | 375
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 41 | 41 | 82
  Georgia | 27 | 33 | 60
  Russia | 89 | 92 | 181
  Ukraine | 43 | 36 | 79
Fertility Status [Count of Participants; unit: Participants]
  of childbearing potential | 59 | 52 | 111
  post menopausal | 120 | 128 | 248
  surgically sterile | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent AEs at Cycle 1
Time Frame: At the end of Cycle 1 (each cycle is 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 200 | 202
Participants | 121 | 122

2. Primary Outcome: Number of Participants With Treatment-emergent AEs All Cycles
Time Frame: At the end of Cycle 4 (each cycle is 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 200 | 202
Participants | 184 | 187

3. Primary Outcome: Number of Participants With Severe (i.e., CTCAE Grade ≥3) TEAEs Reported for ≥2% of Patients in Either Treatment Group and Overall Throughout the Study
Time Frame: At the end of Cycle 4 (each cycle is 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 200 | 202
Participants | 37 | 29

4. Primary Outcome: Number of Participants With Study-Drug-Related TEAEs Reported for ≥2% of Patients in Either Treatment Group Throughout the Study
Time Frame: At the end of Cycle 4 (each cycle is 21 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 200 | 202
Participants | 16 | 22

5. Secondary Outcome: Complete Response in Cycle 1 During the Acute Phase
Description: defined as no emetic episodes [vomit or retch] and no rescue medication
Time Frame: 24 hours after the start of AC chemotherapy administration
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 200 | 202
Participants | 173 | 179

6. Secondary Outcome: Complete Response in Cycle 1 During the Delayed Phase
Description: defined as no emetic episodes [vomit or retch] and no rescue medication
Time Frame: 120 hour after the start of AC chemotherapy administration
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 200 | 202
Participants | 151 | 159

7. Secondary Outcome: Complete Response in Cycle 1 During the Overall Phase
Description: defined as no emetic episodes [vomit or retch] and no rescue medication
Time Frame: 0-120 hours after the start of AC chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 200 | 202
Participants | 146 | 156

8. Secondary Outcome: Overall Percentage of Patients With NIDL Based on FLIE Scores for Cycles 1
Description: Percentage (including two-sided 95% CI using Wilson score method) of patients with NIDL based on FLIE scores (overall, by domain, and by individual item) are summarized by treatment group. NIDL was defined as a score greater than 108 points, 54 points, and 6 points for total FLIE score, domain score, and single item score, respectively. Differences between treatment groups for total FLIE score and domain scores (nausea and vomiting) were presented with two-sided 95% CIs using the CMH method adjusted for region and age class strata and also using Newcombe-Wilson's method without strata adjustment.
  No Impact on Daily Life (NIDL) Based on Functional Living Index-Emesis (FLIE) Scores. The FLIE is a nausea and vomiting specific self report instrument comprised of two domains (nausea and vomiting) with nine identical items in each domain
Time Frame: cycle 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 200 | 202
percentage of participants
  total score | 74.0 [67.5 to 79.6] | 78.7 [72.6 to 83.8]
  Nausea domain score | 67.5 [60.7 to 73.6] | 68.3 [61.7 to 74.3]
  Vomiting domain score | 87.5 [82.2 to 91.4] | 90.6 [85.8 to 93.9]

ADVERSE EVENTS:
Time Frame: from screening (day -14) to end of follow up (Day 22) of Cycle 4
Arm/Group | Test Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/200 | 0/202
Serious Adverse Events (participants affected / at risk) | 5/200 | 4/202
Other Adverse Events (participants affected / at risk) | 184/200 | 187/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Group (N=200) | Control Group (N=202)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Test Group (N=200) | Control Group (N=202)
Leukopenia (Blood and lymphatic system disorders) | 40 | 33
Anaemia (Blood and lymphatic system disorders) | 31 | 24
Neutropenia (Blood and lymphatic system disorders) | 25 | 24
Nausea (Gastrointestinal disorders) | 14 | 9
Diarrhoea (Gastrointestinal disorders) | 10 | 9
Fatigue (General disorders) | 30 | 34
Asthenia (General disorders) | 27 | 17
Gamma-glutamyltransferase increased (Investigations) | 11 | 7
Headache (Nervous system disorders) | 10 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 143 | 138

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT03403712/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT03403712/SAP_001.pdf